CLINICAL TRIAL: NCT03386344
Title: A 26-week Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Phase 3 Study With a 78-week Extension Period to Evaluate the Efficacy and Bone Safety of Sotagliflozin in Patients 55 Years or Older With Type 2 Diabetes Mellitus and Inadequate Glycemic Control
Brief Title: Efficacy and Bone Safety of Sotagliflozin 400 and 200 mg Versus Placebo in Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Acronym: SOTA-BONE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated prematurely for financial reasons and Covid-19 pandemic.
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15294; 2017-002041-30; U1111-1195-6371 (Other: UTN)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Following a 2 week run-in period, participants were randomized to matching placebo to sotagliflozin administered as 2 tablets, once daily, before the first meal of the day, for up to 26 weeks in the Core Treatment Period. Participants were eligible to continue treatment in the Extension Period. The total treatment duration was planned for up to 106 weeks.
  Interventions: Drug: Placebo
- Sotagliflozin 200 mg (Experimental): Following a 2 week run-in period, participants were randomized to Sotagliflozin 200 mg administered as 1 sotagliflozin tablet and 1 matching placebo tablet, once daily, before the first meal of the day, for up to 26 weeks in the Core Treatment Period. Participants were eligible to continue treatment in the Extension Period. The total treatment duration was planned for up to 104 weeks.
  Interventions: Drug: Sotagliflozin; Drug: Placebo
- Sotagliflozin 400 mg (Experimental): Following a 2 week run-in period, participants were randomized to Sotagliflozin 400 mg administered as two 200 mg sotagliflozin tablets, once daily, before the first meal of the day, for up to 26 weeks in the Core Treatment Period. Participants were eligible to continue treatment in the Extension Period. The total treatment duration was planned for up to 104 weeks.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Pharmaceutical form: Tablet; Route of administration: Oral
  Other Names: SAR439954
  Arms: Sotagliflozin 200 mg; Sotagliflozin 400 mg
Drug: Placebo — Pharmaceutical form: Tablet; Route of administration: Oral
  Arms: Placebo; Sotagliflozin 200 mg

SUMMARY:
The primary objective is to demonstrate the superiority of Sotagliflozin 400 milligrams (mg) versus placebo with respect to hemoglobin A1c (Hb1Ac) reduction in participants with type 2 diabetes (T2D) who have inadequate glycemic control on diet and exercise only or with a stable antidiabetes regimen.

DETAILED DESCRIPTION:
Study duration per participant is approximately 110 weeks (Screening period of up to 2 weeks, 2 week single-blind run-in period), a 26-week double-blind core treatment period, a 78-week double-blind extension period, and a 2- week post treatment follow up period.

Dual-energy X-ray absorptiometry (DXA) scans will be performed to assess Bone Mineral Density and Fat vs. Lean body mass at baseline and Weeks 26, 52, and 104.

ELIGIBILITY:
Inclusion criteria :

* Participants with T2D managed with diet and exercise only or with a stable antidiabetes regimen (in monotherapy or combination therapy that can include oral antidiabetes medications, insulin, or glucagon-like peptide-1 agonists) for more than 12 weeks.
* Participants has given written informed consent to participate in the study in accordance with local regulations.

Exclusion criteria:

* Age <55 years.
* Women who have been postmenopausal (or undergone bilateral oophorectomy) for less than 5 years.
* Type 1 diabetes mellitus.
* Body mass index (BMI) ≤20 or >45 kilogram per meter square kg/m^2 or bodyweight that exceeds the weight limits of the DXA scanner.
* Hemoglobin A1C (HbA1c) <7.0% or HbA1c >11.0%.
* Use of a selective sodium-glucose cotransporter type 2 (SGLT2) inhibitor or thiazolidinedione within 24 months.
* Bone mineral density (BMD) T- score <-2.0 at any site (ie, lumbar spine, total hip, or femoral neck).
* History of fracture within 12 months (except for fractures of the hand/fingers, foot/toes, facial bones, and skull).
* Treatment with medications known to affect bone mass or modify the risk of fractures within 36 months (eg, bisphosphonates, selective estrogen receptor modulators, calcitonin, teriparatide, denosumab, strontium ranelate, growth hormone, aromatase inhibitors, androgen deprivation therapy, carbamazepine, phenytoin, and phenobarbital). Use of hormonal replacement that includes systemic or transdermal estrogen or testosterone is excluded unless is stable for at least 24 months prior to Screening.
* Lower extremity complications (such as skin ulcers, infection, osteomyelitis and gangrene) identified during the Screening period, and still requiring treatment at randomization.
* Uncontrolled high blood pressure, severe anemia, severe cardiovascular problems, such as heart failure, active cancer, or other conditions that the Investigator believes with result in a short life expectancy.
* Renal disease as defined by an estimated glomerular filtration rate (eGFR) <30 milliliter per minute (mL/min)/1.73 meter square (m^2) at the Screening Visit by the 4 variable Modification of Diet in Renal Disease equation.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2020-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (53):
- United States (14):
  - Investigational Site Number 8409009, Escondido, California
  - Investigational Site Number 8409010, Greenbrae, California
  - Investigational Site Number 8409005, Walnut Creek, California
  - Investigational Site Number 8409012, Columbus, Georgia
  - Investigational Site Number 8409011, Evansville, Indiana
  - Investigational Site Number 8409014, Wichita, Kansas
  - Investigational Site Number 8409015, Albuquerque, New Mexico
  - Investigational Site Number 8409002, Chapel Hill, North Carolina
  - Investigational Site Number 8409001, Wilmington, North Carolina
  - Investigational Site Number 8409008, Dayton, Ohio
  - Investigational Site Number 8409004, Chattanooga, Tennessee
  - Investigational Site Number 8409013, Austin, Texas
  - Investigational Site Number 8409003, Dallas, Texas
  - Investigational Site Number 8409007, Katy, Texas
- Australia (3):
  - Investigational Site Number 0369003, Fremantle
  - Investigational Site Number 0369002, Merewether
  - Investigational Site Number 0369004, Parkville
- Canada (7):
  - Investigational Site Number 1249003, Brampton
  - Investigational Site Number 1249008, Etobicoke
  - Investigational Site Number 1249005, Pointe-Claire
  - Investigational Site Number 1249006, Thornhill
  - Investigational Site Number 1249004, Thornhill
  - Investigational Site Number 1249007, Vancouver
  - Investigational Site Number 1249002, Victoriaville
- Mexico (6):
  - Investigational Site Number 4849001, Aguascalientes
  - Investigational Site Number 4849006, Aguascalientes, Aguascalientes
  - Investigational Site Number 4849003, Cuernavaca
  - Investigational Site Number 4849002, Guadalajara Jalisco
  - Investigational Site Number 4849004, Monterrey
  - Investigational Site Number 4849005, Xalapa
- New Zealand (4):
  - Investigational Site Number 5549004, Auckland
  - Investigational Site Number 5549003, Christchurch
  - Investigational Site Number 5549001, Rotorua
  - Investigational Site Number 5549002, Wellington
- Russia (6):
  - Investigational Site Number 6439007, Kemerovo
  - Investigational Site Number 6439005, Novosibirsk
  - Investigational Site Number 6439001, Saint Petersburg
  - Investigational Site Number 6439002, Saint Petersburg
  - Investigational Site Number 6439003, Saint Petersburg
  - Investigational Site Number 6439006, Yaroslavl
- South Korea (5):
  - Investigational Site Number 4109006, Daejeon
  - Investigational Site Number 4109005, Guri-Si, Gyeonggi-Do
  - Investigational Site Number 4109003, Gyeonggi-do
  - Investigational Site Number 4109004, Seoul
  - Investigational Site Number 4109001, Seoul
- Taiwan (8):
  - Investigational Site Number 1589005, Changhua
  - Investigational Site Number 1589008, New Taipei City
  - Investigational Site Number 1589006, Taichung
  - Investigational Site Number 1589007, Taichung
  - Investigational Site Number 1589001, Tainan
  - Investigational Site Number 1589002, Tainan
  - Investigational Site Number 1589004, Taipei
  - Investigational Site Number 1589003, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 53 investigative sites in the United States, Australia, Canada, Korea, Republic of Mexico, New Zealand, Russian Federation, and Taiwan from 19 February 2018 to 30 May 2020.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus (DM), were enrolled in 1 of 3 treatment groups: Placebo, Sotagliflozin 200 milligrams (mg) or Sotagliflozin 400 mg.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Started | 126 | 125 | 125
Completed | 9 | 9 | 9
Not Completed | 117 | 116 | 116
Not completed — Adverse Event | 6 | 3 | 1
Not completed — Poor Compliance to Protocol | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 101 | 102 | 106
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — At the Participant's own Request | 7 | 7 | 8
Not completed — Reason not Specified | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The randomized population included any participant who had been allocated to a randomized treatment regardless of whether the treatment kit was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 126 | 125 | 125 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (5.7) | 66.1 (6.7) | 66.5 (6.9) | 66.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 55 | 167
  Male | 70 | 69 | 70 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 21 | 23 | 67
  Not Hispanic or Latino | 102 | 104 | 102 | 308
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3 | 6
  Asian | 26 | 25 | 24 | 75
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3 | 6
  Black or African American | 8 | 8 | 6 | 22
  White | 88 | 87 | 88 | 263
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Austria | 2 | 8 | 3 | 13
  Canada | 20 | 17 | 20 | 57
  South Korea | 8 | 9 | 7 | 24
  Mexico | 16 | 14 | 17 | 47
  New Zealand | 9 | 9 | 11 | 29
  Russia | 17 | 14 | 19 | 50
  Taiwan | 12 | 9 | 7 | 28
  United States | 42 | 45 | 41 | 128
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.38 (0.91) | 8.32 (0.96) | 8.32 (0.95) | 8.34 (0.94)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 133.04 (13.10) | 131.48 (13.69) | 134.65 (14.74) | 133.06 (13.88)
Bone Mineral Density (BMD) T-score: Lumbar Spine [Mean (Standard Deviation); unit: t-score] — BMD T-score Reference Ranges: Score (-1.0 and above): bone density is considered normal; Score (Between -1.0 and -2.5): sign of osteopenia, a condition that may lead to osteoporosis; Score (-2.5 and below): indicates likely osteoporosis.
  t-score | 0.69 (2.0) | 0.70 (1.74) | 0.88 (1.71) | 0.76 (1.82)
BMD T-score: Total Hip [Mean (Standard Deviation); unit: t-score] — BMD T-score Reference Ranges: Score (-1.0 and above): bone density is considered normal; Score (Between -1.0 and -2.5): sign of osteopenia, a condition that may lead to osteoporosis; Score (-2.5 and below): indicates likely osteoporosis.
  t-score | 0.13 (1.01) | 0.00 (0.90) | 0.24 (1.17) | 0.12 (1.04)
BMD T-score: Femoral Neck [Mean (Standard Deviation); unit: t-score] — BMD T-score Reference Ranges: Score (-1.0 and above): bone density is considered normal; Score (Between -1.0 and -2.5): sign of osteopenia, a condition that may lead to osteoporosis; Score (-2.5 and below): indicates likely osteoporosis.
  t-score | -0.69 (0.86) | -0.66 (0.88) | -0.46 (1.03) | -0.60 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 26
Description: An analysis of covariance (ANCOVA) model is used for analysis.
Time Frame: Baseline to Week 26
Population: Intent-to-treat (ITT) population included all randomized participants, irrespective of compliance with the study protocol and procedures. Missing data are imputed using washout imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 126 | 125 | 125
percentage of HbA1c | -0.22 (0.080) | -0.66 (0.077) | -0.67 (0.079)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of sex (male, female), and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares (LS) Means = -0.45, 95% CI 2-sided [-0.649 to -0.250], Standard Error of Mean 0.102
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -0.43, 95% CI 2-sided [-0.634 to -0.235], Standard Error of Mean 0.102

2. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Lumbar Spine at Week 26
Description: An ANCOVA model is used for analysis.
Time Frame: Baseline to Week 26
Population: Safety population included all randomized participants who had received at least one dose of investigational medicinal product (IMP). Missing data are imputed using a pattern-based imputation method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 125 | 125 | 125
percent change | 0.37 (0.327) | 0.13 (0.323) | 0.22 (0.327)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; Percent change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of sex (male, female), and country as fixed effects, and baseline BMD as a covariate; Test type: Superiority; p = 0.5707, ANCOVA; Difference in LS Means = -0.24, 95% CI 2-sided [-1.070 to 0.590], Standard Error of Mean 0.423
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7247, ANCOVA; Difference in LS Means = -0.15, 95% CI 2-sided [-0.969 to 0.674], Standard Error of Mean 0.419

3. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Total Hip at Week 26
Description: An ANCOVA model is used for analysis.
Time Frame: Baseline to Week 26
Population: Safety population included all randomized participants who had received at least one dose of IMP. Missing data are imputed using a pattern-based imputation method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 125 | 125 | 125
percent change | -0.36 (0.259) | -0.22 (0.220) | -0.16 (0.223)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; Percent change from baseline to Week 26 was analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of sex (male, female), and country as fixed effects, and baseline lumbar spine as a covariate; Test type: Superiority; p = 0.6454, ANCOVA; Difference in LS Means = 0.14, 95% CI 2-sided [-0.462 to 0.745], Standard Error of Mean 0.308
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5289, ANCOVA; Difference in LS Means = 0.19, 95% CI 2-sided [-0.410 to 0.798], Standard Error of Mean 0.308

4. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Femoral Neck at Week 26
Description: An ANCOVA model is used for analysis.
Time Frame: Baseline to Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 125 | 125 | 125
percent change | -0.94 (0.379) | -0.20 (0.332) | -0.62 (0.338)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; Percent change from baseline to Week 26 was analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of sex (male, female), and country as fixed effects, and baseline BMD as a covariate; Test type: Superiority; p = 0.1050, ANCOVA; Difference in LS Means = 0.75, 95% CI 2-sided [-0.157 to 1.654], Standard Error of Mean 0.462
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.4804, ANCOVA; Difference in LS Means = 0.32, 95% CI 2-sided [-0.577 to 1.226], Standard Error of Mean 0.460

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: An ANCOVA model is used for analysis.
Time Frame: Baseline to Week 26
Population: ITT population included all randomized participants, irrespective of compliance with the study protocol and procedures. Missing data are imputed using washout imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 126 | 125 | 125
kilogram (kg) | -0.46 (0.261) | -2.37 (0.258) | -2.16 (0.264)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of sex (male, female), and country as fixed effects, and baseline body weight as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -1.91, 95% CI 2-sided [-2.568 to -1.252], Standard Error of Mean 0.336
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -1.70, 95% CI 2-sided [-2.360 to -1.046], Standard Error of Mean 0.335

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: An ANCOVA model is used for analysis.
Time Frame: Baseline to Week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 126 | 125 | 125
milligram per deciliter (mg/dL) | -7.274 (3.6064) | -26.165 (3.4656) | -28.607 (3.5912)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of sex (male, female), and country as fixed effects, baseline fasting plasma glucose as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -18.891, 95% CI 2-sided [-27.8605 to -9.9205], Standard Error of Mean 4.5766
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -21.333, 95% CI 2-sided [-30.3294 to -12.3360], Standard Error of Mean 4.5902

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 12
Description: An ANCOVA model is used for analysis.
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 126 | 125 | 125
millimeter of mercury (mmHg) | -0.80 (1.149) | -1.61 (1.130) | -1.97 (1.165)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 12 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of sex (male, female), and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.5864, ANCOVA; Difference in LS Means = -0.80, 95% CI 2-sided [-3.705 to 2.095], Standard Error of Mean 1.480
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.4315, ANCOVA; Difference in LS Means = -1.16, 95% CI 2-sided [-4.058 to 1.734], Standard Error of Mean 1.478

8. Secondary Outcome: Percentage of Participants With Hemoglobin A1c (HbA1c) <7.0% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants, irrespective of compliance with the study protocol and procedures.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 126 | 125 | 125
percentage of participants | 9.5 | 20.0 | 21.6
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; Percentage difference between treatment groups from randomization strata of HbA1c (≤8.5, >8.5%) at screening and randomization strata of sex (male, female) using Cochran-Mantel-Haenszel weights; Test type: Superiority; p = 0.0172, Cochran-Mantel-Haenszel; Percentage Difference = 10.5, 95% CI 2-sided [1.78 to 19.23]
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0076, Cochran-Mantel-Haenszel; Percentage Difference = 12.0, 95% CI 2-sided [3.23 to 20.86]

9. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Time Frame: up to 106 weeks
Population: Safety population included all randomized participants who had received at least one dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 125 | 125 | 125
percentage of participants | 80.0 | 82.4 | 82.4

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose of study drug (up to 104 weeks) + 2 weeks
Description: The safety population included all randomized participants who had received at least one dose of IMP.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 1/125 | 0/125 | 0/125
Serious Adverse Events (participants affected / at risk) | 20/125 | 10/125 | 9/125
Other Adverse Events (participants affected / at risk) | 66/125 | 67/125 | 68/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=125) | Sotagliflozin 200 mg (N=125) | Sotagliflozin 400 mg (N=125)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Maisonneuve fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=125) | Sotagliflozin 200 mg (N=125) | Sotagliflozin 400 mg (N=125)
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 16
Influenza (Infections and infestations) | 2 | 11 | 5
Nasopharyngitis (Infections and infestations) | 12 | 9 | 11
Upper respiratory tract infection (Infections and infestations) | 24 | 15 | 3
Urinary tract infection (Infections and infestations) | 15 | 11 | 14
Fall (Injury, poisoning and procedural complications) | 9 | 4 | 7
Bone density decreased (Investigations) | 5 | 10 | 7
Vitamin D deficiency (Metabolism and nutrition disorders) | 9 | 12 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 5 | 5
Headache (Nervous system disorders) | 8 | 3 | 5
Pollakiuria (Renal and urinary disorders) | 1 | 7 | 3
Hypertension (Vascular disorders) | 7 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03386344/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT03386344/SAP_001.pdf